CLINICAL TRIAL: NCT04435158
Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity Study Following Multiple Subcutaneous Injections of SHR-1222 in Postmenopausal Osteoporosis Patients
Brief Title: A Multiple Dose Study to Evaluate the Effect of SHR-1222 Injection in Postmenopausal Osteoporosis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1222-102
Record Dates: First submitted 2020-06-11; First posted 2020-06-17 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1：SHR-1222 (Experimental): Subcutaneous injection of SHR-1222 dosage 1 monthly × 6 months
  Interventions: Drug: SHR-1222
- Cohort 2：SHR-1222 (Experimental): Subcutaneous injection of SHR-1222 dosage 2 monthly × 6 months
  Interventions: Drug: SHR-1222
- Cohort 3：SHR-1222 (Experimental): Subcutaneous injection of SHR-1222 dosage 3 monthly × 6 months
  Interventions: Drug: SHR-1222
- Cohort 4：SHR-1222 (Experimental): Subcutaneous injection of SHR-1222 dosage 4 every 2 months × 6 months
  Interventions: Drug: SHR-1222
- Cohort 5：SHR-1222 (Experimental): Subcutaneous injection of SHR-1222 dosage 5 every 2 months × 6 months
  Interventions: Drug: SHR-1222
- Cohort 6：placebo (Experimental): Subcutaneous injection of placebo × 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1222 — Pharmaceutical form: water injection Route of administration: subcutaneous injection
  Arms: Cohort 1：SHR-1222; Cohort 2：SHR-1222; Cohort 3：SHR-1222; Cohort 4：SHR-1222; Cohort 5：SHR-1222
Drug: Placebo — Pharmaceutical form: water injection Route of administration: subcutaneous injection
  Arms: Cohort 6：placebo

SUMMARY:
This is a Multi-Center, Randomized, Double-Blind, Dose Escalation, Placebo Parallel Controlled PhaseⅠClinical study to Evaluate the Safety, Tolerability and Pharmacokinetics, Pharmacodynamics, Immunogenicity with Multiple Subcutaneous Injections of SHR-1222 in Postmenopausal Osteoporosis Patients.

The primary objective of this study is to investigate the safety and tolerability of a range of subcutaneous SHR-1222 in postmenopausal osteoporosis patients. Secondary objectives are to determine the pharmacokinetics (PK), pharmacodynamics (PD) profile of SHR-1222 in postmenopausal osteoporosis patients including assessment of immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. Age ≥50 and ≤70 years old and post menopause for at least 5 years at the time of screening;
3. Weight ≥40kg at the time of screening;
4. BMD T-score ≤ -2.50 at the lumbar vertebrae, total hip or femoral neck at the time of screening, based on DXA scans;
5. At least 2 vertebrae in the L1-L4 region and at least one hip are evaluable by DXA;
6. Without disease that would significantly affect the study or bring additional health risks at the time of screening or baseline; blood pressure < 150 / 95mmHg, blood fasting blood glucose < 7.0mmol/l, glycosylated hemoglobin < 7%, or total cholesterol < 6.2mmol/l, triglyceride < 3.4mmol/l under the condition of lifestyle improvement rather than drug treatment; If there are other abnormalities in the examination report of the subject, the subject could only be included after investigator approval;
7. Ambulatory.

Exclusion Criteria:

1. Any disease affecting bone metabolism;
2. Any severe (SQ3) or more than 2 moderate (SQ2) vertebral fractures, as assessed by the central imaging based on lateral spine x-rays at the time of screening;
3. History of hip fracture;
4. 25 (OH) vitamin D levels < 20 ng/mL at the time of screening. Vitamin D repletion will be permitted and subjects may be rescreened;
5. BMD T-score < -3.50 at the lumber vertebra, total hip or femoral neck at the time of screening, based on DXA scans;
6. Use of the following agents affecting bone metabolism:

   * IV bisphosphonates or denosumab prior to screening;
   * Oral bisphosphonates, PTH analogs, Strontium or fluoride within 12m prior to screening;
   * Hormone replacement therapy within 6m prior to screening;
   * Glucocorticosteroids (inhaled or topical corticosteroids administered more than 2 weeks before the enrollment date are allowed), Anabolic steroids, Calcitriol and available analogues, thiazide diuretics within 3m prior to screening;
7. History of metabolic or bone disease (except osteoporosis) that may interfere with the interpretation of the results, such as hyperprolactinemia, osteosclerosis, Paget's disease, rheumatoid arthritis, osteomalacia, osteogenesis imperfecta, osteopetrosis, ankylosing spondylitis, Cushing's disease, hyperprolactinemia, and malabsorption syndrome;
8. Hyperparathyroidism, hypothyroidism, hyperthyroidism, hypothyroidism, hypercalcemia, hypocalcemia, renal failure, etc at the time of screening;
9. Malignancy except non-melanoma skin cancers, cervical or breast ductal carcinoma in situ within the last 5 years;
10. A clinical history of drug allergy or a history of atopic allergic diseases (asthma, urticaria, eczema dermatitis) or a known allergy to experimental or similar experimental drugs;
11. Past medical history of cerebral infarction, ischemic or hemorrhagic stroke;
12. Past medical history of Myocardial infarction, coronary heart disease, angina pectoris, heart failure (cardiac function II-IV), serious arrhythmia (such as atrial fibrillation, pacemaker needed)
13. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or gamma pancreatic acyl transferase (GGT) or total bilirubin, more than 2 x ULN during screening;
14. 3 months prior to screening involved in any drug clinical subjects (except screening failed or not given cinical drugs) or within 5 half-lives of test drug at the time of screening;
15. Any major surgery in 1m prior to screening or a surgery plan during the study;
16. Blood donation or loss more than 400mL or blood transfusion within 3 months prior to screening;
17. Human immunodeficiency virus antibody (HIV-ab), syphilis serological examination, hepatitis b virus surface antigen (HBsAg), hepatitis c virus antibody (HCV-ab) were positive;
18. No history of alcohol and substance abuse or positive urine drug screening;
19. Subjects with any other situation should not be involved, which determined by the researchers.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerance: Number of subjects with adverse events | Dose administration to 225 days after first dose administration
  Number & proportion of subjects with adverse events

SECONDARY OUTCOMES:
Assessment of PK parameter-time to maximum concentration (Tmax) | Pre-dose to 225 days after first dose administration
Assessment of PK parameter-maximum concentration (Cmax) | Pre-dose to 225 days after first dose administration
Assessment of PK parameter-area under curve (AUC) | Pre-dose to 225 days after first dose administration
Assessment of PD parameter-change in serum C-telopeptide (sCTx) from baseline | Pre-dose to 225 days after first dose administration
Assessment of PD parameter-change in aminoterminal propeptide type-1 procollagen (P1NP) from baseline | Pre-dose to 225 days after first dose administration
Assessment of PD parameter-change in osteocalcin from baseline | Pre-dose to 225 days after first dose administration
Assessment of PD parameter-change in bone-specific alkaline phosphatase (BSAP) from baseline | Pre-dose to 225 days after first dose administration
Assessment of PD parameter-change in serum totol sclerostin | Pre-dose to 225 days after first dose administration
Assessment of PD parameter-change in areal bone mineral density of lumbar spine (L1-L4) from baseline by dualenergy X-ray absorptiometry | Pre-dose to 225 days after first dose administration
Assessment of PD parameter-change in areal bone mineral density of collum femoris from baseline by dualenergy X-ray absorptiometry | Pre-dose to 225 days after first dose administration
Assessment of PD parameter-change in areal bone mineral density of total hip from baseline by dualenergy X-ray absorptiometry | Pre-dose to 225 days after first dose administration
Antidrug antibody | Pre-dose to 225 days after first dose administration
Neutralizing Antibody | Pre-dose to 225 days after first dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguang Zhou, Principal Investigator — 2nd Xiangya Hospital of Central South University
Locations (1):
- 2nd Xiangya Hospital , Chinese Academy of Medical Sciences, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided